CLINICAL TRIAL: NCT04904289
Title: Early Recognition and Dynamic Risk Warning System of Multiple Organ Dysfunction Syndrome Caused by Sepsis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wu Jianfeng, prof, Sun Yat-sen University
Other Study IDs: Early recognized of MODS
Record Dates: First submitted 2021-05-23; First posted 2021-05-27 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Sepsis; MODS
Keywords: Sepsis; MODS; Big data; Artificial intelligence
MeSH Terms: conditions — Sepsis; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum, Urine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis with MODS: Patients with sepsis occurred MODS.
  Interventions: Other: All intervention of real world
- Sepsis without MODS: Patients with sepsis did not occur MODS.
  Interventions: Other: All intervention of real world

INTERVENTIONS:
Other: All intervention of real world — We analyzed all data we can obtain from our databases

SUMMARY:
Background Sepsis still the main challenge of ICU patients, because of its high morbidity and mortality. The proportion of sepsis, severe sepsis, and septic shock in china were 3.10%, 43.6%, and 53.3% with a 2.78%, 17.69%, and 51.94%, of 90-day mortality, respectively.

Besides, according to the latest definition of sepsis- "a life-threatening organ dysfunction caused by a dysregulated host response to infection. ", it is a disease with intrinsic heterogeneity. Sepsis as a syndrome with such great heterogeneity, there will be significant differences in the severity of sepsis. As a result, there will be significant differences in the treatment and monitoring intensity required by patients with severe sepsis and mild sepsis. No matter from the economic perspective or from the risk of treatment, a proper level of treatment will be the best chose of patient. However, the evaluation of the sepsis severity was not satisfied. Such of SOFA, the AUC of predict patients' mortality was only 69%. Weather these patients occurred multiple organ dysfunction syndrome (MODS) may had totally different outcome and needed totally different treatment. All these treatments need early interference, in order to achieve a good prognosis. Hence, early recognition of MODS caused by sepsis became an imperious demand.

Study design On the base of regional critical medicine clinical information platform, a multi-center, sepsis big data platform (including clinical information database and biological sample database) and a long-term follow-up database will be established. Thereafter, an early identification, risk classification and dynamic early warning system of sepsis induced MODS will be established. This system was based on the real-time dynamic vital signs and clinical information, combined with biomarker and multi-omics information. And this system was evaluated sepsis patients via artificial intelligence, machine learning, bioinformatics analysis techniques.

Finally, optimize the early diagnosis of sepsis induced MODS, standardized the treatment strategy, reduce the morbidity and mortality of MODS through this system.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with sepsis3.0

Exclusion Criteria:

* Patients' data missing is greater than 20%

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis
Sampling Method: Probability Sample
Enrollment: 60000 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the MODS recognized system | 90 days
Specificity of the MODS recognized system | 90 days
The AUC of the MODS recognized system ROC | 90 days

SECONDARY OUTCOMES:
The Incidence rate of MODS in sepsis patients | 90 days
  The Incidence rate of MODS in Chinese sepsis patients
The mortality of MODS in sepsis patients | 90 days
  The mortality of MODS in Chinese sepsis patients

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing General Hospital of Nanjing Military Commend, Nanjing, Jiangsu
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Beijing Friendship Hospital, Capital Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xie J, Wang H, Kang Y, Zhou L, Liu Z, Qin B, Ma X, Cao X, Chen D, Lu W, Yao C, Yu K, Yao X, Shang H, Qiu H, Yang Y; CHinese Epidemiological Study of Sepsis (CHESS) Study Investigators. The Epidemiology of Sepsis in Chinese ICUs: A National Cross-Sectional Survey. Crit Care Med. 2020 Mar;48(3):e209-e218. doi: 10.1097/CCM.0000000000004155. PMID 31804299
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Stanski NL, Wong HR. Prognostic and predictive enrichment in sepsis. Nat Rev Nephrol. 2020 Jan;16(1):20-31. doi: 10.1038/s41581-019-0199-3. Epub 2019 Sep 11. PMID 31511662
- [Background] Liu Z, Meng Z, Li Y, Zhao J, Wu S, Gou S, Wu H. Prognostic accuracy of the serum lactate level, the SOFA score and the qSOFA score for mortality among adults with Sepsis. Scand J Trauma Resusc Emerg Med. 2019 Apr 30;27(1):51. doi: 10.1186/s13049-019-0609-3. PMID 31039813